CLINICAL TRIAL: NCT02759978
Title: Individualized Diagnosis of Endocarditis and Its Therapy With a Focus on Infected Prosthetic materiAL
Acronym: IDENTICAL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Bhanu Sinha, MD, PhD, Principal Investigator, University Medical Center Groningen
Other Study IDs: M16.189348
Record Dates: First submitted 2016-04-18; First posted 2016-05-03 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Endocarditis; Prosthetic Material Related Infection
Keywords: Imaging; Computed Tomography; Magnetic Resonance Imaging; Positron Emission Tomography; Leukocyte Scintigraphy; Microbiological diagnostics; Sonication; Drug Monitoring; Cardiac Surgery
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Suspicion NVE: Patients with suspicion of native valve endocarditis, infective endocarditis and no intracardiac prosthetic material in situ
  Interventions: Other: diagnostic workup
- Suspicion (PVE): Patients with a suspicion of prosthetic valve endocarditis (PVE), infective endocarditis and one or more prosthetic valves in situ
  Interventions: Other: diagnostic workup
- Suspicion pacemaker/ICD related endocarditis: Patients with a suspicion of infective endocarditis and a pacemaker or implantable cardiac defibrillator (ICD) in situ
  Interventions: Other: diagnostic workup

INTERVENTIONS:
Other: diagnostic workup — Our primary objective is to test whether the proportion of patients diagnosed correctly with the use of 18F-FDG-PET/CT, MD-CTA, and 18F-FDG-PET/MD-CTA added to the gold standard in current clinical practice, the modified Duke criteria by Li et al. 2000, is significantly higher as compared with the modified Duke criteria on itself. The gold standard is clinical judgement after clinical follow-up by a multidisciplinary team with medical specialists.

SUMMARY:
Infective endocarditis (IE) is a frequent and serious complication of implanted intracardiac prosthetic material, with a high morbidity and mortality. Therefore, this study aims to improve outcome of IE, with a focus on patients with intracardiac prosthetic material. In this study the investigators deal with research questions about both the diagnosis (microbiological, imaging, and expert opinion) and treatment of IE (with antimicrobial agents and surgical), in order to improve these clinical components and ultimately aim to improve outcome.

DETAILED DESCRIPTION:
Rationale

Infective endocarditis (IE) is a frequent and serious complication of implanted intracardiac prosthetic material, with a high morbidity and mortality. The number of procedures where prosthetic material is implanted in the heart increases, as do the age and comorbidity of treated subjects. In current clinical practice diagnosis of infected intracardiac prosthetic material is often difficult because of the lack of sensitivity of the available diagnostic armamentarium for IE.

As a general rule, first line treatment of intracardiac prosthetic material related endocarditis consists of surgical prosthesis removal, combined with appropriate antimicrobial therapy. The exception encompasses uncomplicated prosthetic valve endocarditis (PVE). PVE actually has a fair chance of successful medical treatment alone (>50%), depending on the causative micro-organism. Although there is evidence and consensus with regard to the first line treatment, surgical removal is not always possible because of its associated high risk, technical limitations, or unwillingness of patients to undergo an invasive surgical procedure. Second and third line treatments do not include surgery, and consist of antimicrobial therapy with biofilm-penetrating agents during a predetermined timespan (second line) or as life-long suppressive antimicrobial therapy (third line). These treatments are the alternative in situations wherein first line treatment is not feasible or is unwanted. Although not extensively investigated, these treatments are considered suboptimal.

Therefore further research is necessary. More research is needed to diagnose IE more accurate and prompt, as current diagnostic criteria (the modified Duke criteria) for IE are insufficient and as it is unclear how to best allocate non-invasive imaging techniques, especially for intracardiac prosthetic material. More research is also needed to verify the indications for and optimize the use of second and third line treatments in patients with intracardiac prosthetic material.

Objectives

Primary

To define the diagnostic value of the combination of 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose positron emission tomography (18F-FDG PET) and electrocardiogram-gated multidetector computed tomography angiography (ECG-gated MD-CTA) in patients suspected of IE, in particular those with intracardiac prosthetic material, when added to the standard diagnostic work-up for IE.

Secondary

* To define the predictive value of MD-CTA and 18F-FDG PET with regard to relapse rate and mortality of IE;
* To identify sources of false positive and false negative results in MD-CTA and 18F-FDG PET (e.g. the effect of the use of antimicrobial therapy on imaging findings);
* To identify the best MD-CTA and 18F-FDG PET scanning protocol;
* To define the role of 18F-FDG PET for finding other infectious lesions in the body;
* To assess and compare current clinical practices in patients with intracardiac prosthetic material related infection when the foreign material cannot be removed; to determine the outcomes of second and third line treatment as compared with first line treatment, and to determine predictors of outcome;
* To investigate the potential of therapeutic drug monitoring (TDM) to improve the antimicrobial therapy in patients suspected of IE, in particular those with intracardiac prosthetic material:

  * for which peak and through blood concentrations should be aimed at in IE for flucloxacillin, rifampicin, cefazolin, cefuroxime, ceftriaxone, amoxicillin, penicillin; fluconazole, flucytosine, amphotericin-B?
  * for which peak blood concentrations should be aimed at for gentamicin in IE?
  * for which peak and through blood concentrations should be aimed at for vancomycin in intracardiac prosthetic material related IE?
  * for which through blood concentrations should be aimed at in IE for voriconazole?
* To investigate antimicrobial concentrations in resected cardiac tissue (e.g. heart valve or vegetation which has been removed based on medical indication) in patients with IE who have been treated medically with antimicrobials and who subsequently are operated upon.

Study design

Prospective multicentre observation study, with the University Medical Center Groningen (UMCG) in Groningen as the leading centre.

Study population

Patients (≥18 years) in which IE is suspected according to the britisch society for antimicrobial chemotherapy (BSAC) criteria 2012.

Main study parameters/endpoints

Number of clinically identified (prosthetic material related) endocarditis episodes, according to (multiple) constellation(s) of diagnostic criteria versus number of "true" (prosthetic material related) endocarditis episodes, according to our gold standard "expert opinion after 12 months (+/- 2 weeks) follow-up" (based on clinical reasoning, the modified Duke criteria, and findings during surgery and from pathology).

ELIGIBILITY:
Inclusion Criteria:

* patients presenting to participating hospitals
* age ≥18 years
* BSAC-criteria 2012: suspicion of infective endocarditis, retained in the differential diagnosis after clinical reasoning, without alternative diagnosis

Exclusion Criteria:

* not fulfilling inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (≥18 years) in which infective endocarditis is suspected according to the BSAC-criteria 2012
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-05; Primary Completion 2023-04 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
IE clinical diagnosis | 2 months
  Number of clinically identified (prosthetic material related) endocarditis episodes, according to (multiple) constellation(s) of diagnostic criteria (the current gold standard of the modified Duke criteria, and newly set-up and to be investigated constellations of diagnostic elements)
IE final diagnosis | 1 year
  Number of "true" prosthetic material related endocarditis episodes, according to expert opinion after follow-up (important components being findings during surgery and from pathology)
Relapse/recurrence | 1 year
  Number of relapses / recurrences
1 year mortality | 1 year
  Mortality after 1-year follow-up
30 day mortality | 30 days
  Mortality after 30-days follow-up
Duration of antimicrobial therapy | 30 days
  Duration of antimicrobial therapy (including appropriateness of drug, dosing and dosing regimen)
Cardiac surgery | 1 year
  Cardiac surgery performed
Complications | 1 year
  Number of complications: congestive heart failure (CHF) or other hemodynamic consequences, septic emboli, metastatic infection

SECONDARY OUTCOMES:
Adverse events | 1 year
  Number of adverse and serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bhanu Sinha, MD, PhD, Principal Investigator — Medical Microbiology, University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Currently single center study